CLINICAL TRIAL: NCT00507299
Title: A Safe Environment for Every Kid (SEEK) I: Preventing Child Maltreatment - A Role for Pediatrics
Brief Title: A Safe Environment for Every Kid (SEEK) I
Acronym: SEEK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Howard Dubowitz, Professor of Pediatrics, University of Maryland, Baltimore
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-20890
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2019-11

CONDITIONS: Child Abuse
Keywords: Child maltreatment; Physician education; Prevention

STUDY DESIGN:
Intervention Model Description: Pediatric residents were trained to screen for and help address prevalent psychosocial problems, such as parental depression and substance abuse, that are risk factors for child maltreatment (CM). The SEEK model included a project social worker and use of community resources.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Model Care (SEEK) (Experimental): Residents in this group received special training on addressing pyschosocial problems. They then used a parent screening questionnaire, and addressed identified problems. A study social worker was also part of this intervention. Thus, this group provided enhanced pediatric primary care.
  Interventions: Behavioral: Enhanced pediatric primary care
- Standard pediatric primary care (Active Comparator): This arm involved residents receiving the regular education through the program. They did not use the screening questionnaire to identify psychosocial problems, and did not have a dedicated social worker to assist them. Instead, residents in this group provided standard pediatric primary care
  Interventions: Behavioral: Standard pediatric primary care

INTERVENTIONS:
Behavioral: Enhanced pediatric primary care — Residents received special training to address targeted psychosocial problems. Parents bringing in children (0 - 5 years) completed a screening questionnaire and gave this to their doctor. The resident briefly assessed the identified problems and helped address them. A social worker was present to assist.
  Arms: Model Care (SEEK)
Behavioral: Standard pediatric primary care — Residents did not receive special training on the targeted psychosocial problems. They did not use the parent screening questionnaire, and they did not have a dedicated social worker.
  Arms: Standard pediatric primary care

SUMMARY:
This study aims to enhance pediatric primary care to make it more responsive to psychosocial needs facing many families. We hypothesized that by identifying and addressing certain problems, such as depressed mothers, parental drug use, and domestic violence, we would help decrease child abuse and neglect.

DETAILED DESCRIPTION:
This study aims to enhance pediatric primary care to make it more responsive to psychosocial needs facing many families. We hypothesized that by identifying and addressing certain problems, such as depressed mothers, parental drug use, and domestic violence, we would help decrease child abuse and neglect.

The first step was to train pediatric residents on the importance of addressing the targeted problems. Then, we developed a brief screening tool to use when children under six years came in for the regular checkups. Parents would complete this while waiting for their doctor. Finally, the doctor and/or social worker would try address any problems the parent identified.

ELIGIBILITY:
Inclusion Criteria:

* Child 0 - 5 years
* Family English speaking
* Parent agrees to participate

Exclusion Criteria:

* Child in foster care
* Another child in the family already enrolled

Ages: 1 Month to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2002-06 (Actual); Primary Completion 2005-12-31 (Actual); Study Completion 2006-12-31 (Actual)

PRIMARY OUTCOMES:
Reduced child abuse and neglect | 2002 - 2005
  Reports to Child Protective Services

SECONDARY OUTCOMES:
Improved resident attitudes and behavior regarding psychosocial problems. | 2002 - 2005
  Self-reported thinking and behavior regarding addressing targeted problems

CONTACTS AND LOCATIONS:
Overall Officials: Howard Dubowitz, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Result] Dubowitz H, Feigelman S, Lane W, Prescott L, Blackman K, Grube L, Meyer W, Tracy JK. Screening for depression in an urban pediatric primary care clinic. Pediatrics. 2007 Mar;119(3):435-43. doi: 10.1542/peds.2006-2010. PMID 17332195
- [Derived] Kalra N, Hooker L, Reisenhofer S, Di Tanna GL, Garcia-Moreno C. Training healthcare providers to respond to intimate partner violence against women. Cochrane Database Syst Rev. 2021 May 31;5(5):CD012423. doi: 10.1002/14651858.CD012423.pub2. PMID 34057734
- [Derived] Feigelman S, Dubowitz H, Lane W, Grube L, Kim J. Training pediatric residents in a primary care clinic to help address psychosocial problems and prevent child maltreatment. Acad Pediatr. 2011 Nov-Dec;11(6):474-80. doi: 10.1016/j.acap.2011.07.005. Epub 2011 Sep 29. PMID 21959095